CLINICAL TRIAL: NCT05469633
Title: Application of Portable Ultrasonic Evaluation of Gastric Contents in Painless Gastroscopy
Status: Completed | Type: Observational
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ultrasound and contents
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2022-09

CONDITIONS: Ultrasound Evaluation of Gastric Contents
Keywords: gastric ultrasound; gastric contents; painless electronic gastroscope

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the correlation between gastric ultrasound evaluation and gastroscopic direct vision evaluation of gastric contents, so as to more accurately use gastric ultrasound to evaluate the gastric contents of patients undergoing painless electronic gastroscopy in the outpatient department, so as to develop an individual painless diagnosis and treatment strategy to reduce the risk of lung aspiration.

ELIGIBILITY:
Inclusion Criteria:

* ≥18years
* Patients undergoing painless electronic gastroscopy.
* Voluntarily participate and sign informed consent.

Exclusion Criteria:

* Patients undergoing general electronic gastroscopy.
* Patients who refused to undergo gastric ultrasound.
* Patients with postural difficulties during gastric ultrasonography.
* with fresh wounds or infections at the site of Gastric ultrasound
* Patients whose ultrsound image quality is too poor to properly display the relevant anatomical structures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients undergoing painless electronic gastroscopy were fasted for 8 hours in acccordance with gastroscopy guidelines
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
The cross-sectional area of the antrum (CSA) | Before the painless electronic gastroscopy
  The maximum anteroposterior diameter (recorded as D1) and maximum craniocaudal diameter (recorded as D2) between the gastric antrum serosal surfaces were measured perpendicularly to each other.CSA(cm2) = (π × D1 × D2) / 4
Predicted volume | Before the painless electronic gastroscopy
  Predicted volume calculated by CSA
Observed volume | Before the painless electronic gastroscopy
  All gastric fluid was thoroughly suctioned through an endoscope side port, measured to the nearest mL and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yupei, Study Director — Department of Anesthesiology,The Second Affiliated Hospital ,Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China